CLINICAL TRIAL: NCT05589935
Title: Radicle Relief 1™: A Randomized, Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Pain and Other Health Outcomes
Brief Title: Radicle Relief 1: A Study of Health and Wellness Products on Pain and Other Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-22D05
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pain; Nociceptive Pain; Neuropathic Pain
MeSH Terms: conditions — Pain; Nociceptive Pain; Neuralgia

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control 1 (Placebo Comparator): Relief Product Form 1 - control
  Interventions: Dietary Supplement: Relief Study Product Usage
- Active Product 1.1 (Experimental): Relief Product Form 1 - active product 1
  Interventions: Dietary Supplement: Relief Study Product Usage

INTERVENTIONS:
Dietary Supplement: Relief Study Product Usage — Participants instructed to use study product daily as directed for a period of 4 weeks

SUMMARY:
A randomized, blinded, placebo-controlled study assessing the impact of health and wellness products on pain and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with up to 300 adult participants per study arm, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for less pain, (2) indicate an interest in taking a health and wellness product to potentially help relieve their pain, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data are collected electronically from eligible participants over 5 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses pain as a primary issue (desire for less pain)
* Selects their desire for less pain and/or reduce reliance on medications as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid physical shipping address
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Lack of reliable daily access to the internet
* Reports taking anticoagulants, any medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, or MAOIs
* Reports current or recent (within 3 months) use of chemotherapy, immunotherapy, or oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Change in pain interference | 4 weeks
  Mean difference in pain interference score as assessed by Patient Reported Outcome Measurement System (PROMIS) Pain Interference 6A [scale 6-30; with higher scores corresponding to greater pain interference]

SECONDARY OUTCOMES:
Change in neuropathic pain | 4 weeks
  Mean difference in neuropathic pain score as assessed by PROMIS Neuropathic Pain 5A [scale 5-25; with higher scores corresponding to greater neuropathic pain]
Change in nociceptive pain | 4 weeks
  Mean difference in nociceptive pain score as assessed by PROMIS Nociceptive Pain 5A [scale 5-25; with higher scores corresponding to greater nociceptive pain]
Change in pain intensity | 4 weeks
  Mean difference in pain intensity score as assessed by PROMIS Pain Intensity 1A [scale 1-10; with 0 being 'No pain' and 10 being 'The worst imaginable pain']
Change in feelings of anxiety | 4 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A [scale 4-20; with higher scores corresponding to more severe anxiety]
Change in sleep disturbance | 4 weeks
  Mean difference in sleep disturbance score as assessed by PROMIS Sleep Disturbance Form 4A [scale 4-20; with higher scores corresponding to more severe sleep disturbance]
Minimal clinically important difference (MCID) in pain interference | 4 weeks
  Likelihood of experiencing MCID in pain interference score as assessed by PROMIS Pain Interference 6A
Minimal clinically important difference (MCID) in neuropathic pain | 4 weeks
  Likelihood of experiencing MCID in neuropathic pain score as assessed by PROMIS Neuropathic Pain 5A
Minimal clinically important difference (MCID) in nociceptive pain | 4 weeks
  Likelihood of experiencing MCID in nociceptive pain score as assessed by PROMIS Nociceptive Pain 5A
Minimal clinically important difference (MCID) in pain intensity | 4 weeks
  Likelihood of experiencing MCID in pain intensity score as assessed by PROMIS Pain Intensity 1A

OTHER OUTCOMES:
Change in energy (fatigue) | 4 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 4A [scale 4-20; with higher scores corresponding to greater fatigue]
Change in cognitive function | 4 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognitive Function 4A [scale 4-20; with higher scores corresponding to greater cognitive function]
Change in emotional distress | 4 weeks
  Mean difference in emotional distress score as assessed by PROMIS Emotional Distress- Depression 4A [scale 4-20; with higher scores corresponding to greater levels of emotional distress]
Change in sexual interest | 4 weeks
  Mean difference in sexual interest as assessed by PROMIS Sexual Interest 2.0 [scale 2-10; with higher scores corresponding to greater interest in sexual activity]

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com